CLINICAL TRIAL: NCT04537143
Title: Understanding Imaging Biomarkers That Predict the Progression of Age-Related Macular Degeneration on Multi-modal Novel Retinal Technologies
Brief Title: Image Biomarkers for Progression of AMD
Acronym: IBPAMD
Status: Withdrawn | Type: Observational
Why Stopped: Funding for staff no longer available
Sponsor: Doheny Image Reading Center (Other)
Responsible Party: Principal Investigator, Kenneth Marion, Program Manager - Research, Doheny Image Reading Center
Other Study IDs: Narcisa
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: AMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Non-AMD eyes
- AMD: AMD eyes

SUMMARY:
To study qualitatively and quantitatively the Imaging Biomarkers (IBs) on Multi-modal Imaging with Novel technologies (MINT), in order to understand their role in prediction of the Age-related Macular Degeneration (AMD) progression in eyes with and without treatment. The understanding of IBs will allow early detection of AMD, prediction of its evolution, and guidance for the best options for stratified/individualized treatment of AMD.

DETAILED DESCRIPTION:
The qualitative studies will explore use of OCT Angiography (OCTA), Swept Source OCT (SS-OCT), Ultra-Wide Field Fluorescein Angiography (UWF-FA), Adaptive Optic Scanning Laser Ophthalmoscopy (AO-SLO), Fluorescence Lifetime Imaging Ophthalmoscopy (FLIO), Retro Mode Imaging (RMI) and other novel technologies for the retinal diagnosis. Morphologic qualitative IBs described in the literature like macular neovascularization pattern, retinal tubulations, choriocapillary preservation, retinal pigment epithelium atrophy, drusen patterns, etc as well as other IBPAMD original IBs classified in morphopathogenic categories like IBs related-to-MNV, IBs related-to-atrophy, IBs related-to macular chorio-retinal architecture, etc are analyzed in granular fashion by multi-modal imaging approach before and after different treatments for AMD.

The quantitative IBs assessment will be done in dual mode - classic and original to the IBPAMD trial. The lesions are quantitatively assessed on one hand, by using the classic measurements of the greatest diameter, total lesions area, vessels density, fractal dimension, etc, based on the classic concept of measurements expressed in absolute values (mm, mm2 or pixels). The same lesions are quantitatively assessed by using the original IBPAMD algorithm and software (SITE-app) that introduce a new concept in the quantification of the retinal lesions, the assessment of differences reported to the baseline.

ELIGIBILITY:
Inclusion Criteria:

* being male or female
* at least 18 years of age
* varied ethnic backgrounds (different ethnic groups have different structures of eye anatomy and we must be able to make ethnic subgroups to account for these differences)

Exclusion Criteria:

* vulnerable patients
* patients under 18
* pregnant (we exclude pregnant women because pregnancy often can alter eye anatomy)
* economically and educationally disadvantaged
* decision impaired
* homeless people.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Half control, half AMD eyes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
ONH diameter | 1-2 year FU
area of MNV | 1-2 year FU

IPD SHARING:
Plan to Share IPD: No